CLINICAL TRIAL: NCT05813301
Title: Early Predictors of NAFLD in Patient of Hypothyroidism
Brief Title: NAFLD in Patient of Hypothyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Sawerss Fathy Mihany, Assistant Lecturers, Assiut University
Other Study IDs: NAFLD in Patient of hypothyroi
Record Dates: First submitted 2023-01-13; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most important chronic liver disease in the western world, affecting almost 30% of the general population. Moreover, the prevalence of NAFLD can be higher in type 2 diabetic patients and obese patients, affecting up to 90% of people with a body mass index higher than 40 kg/m2. NAFLD is also the most rapidly increasing cause of hepatic cirrhosis requiring hepatic transplantation in the future. The pathophysiology of NAFLD is complex and involves multiple hits, but the principal contributing factor to its development is hepatic lipid accumulation, which leads to hepatic insulin resistance

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most important chronic liver disease in the western world, affecting almost 30% of the general population. Moreover, the prevalence of NAFLD can be higher in type 2 diabetic patients and obese patients, affecting up to 90% of people with a body mass index higher than 40 kg/m2. NAFLD is also the most rapidly increasing cause of hepatic cirrhosis requiring hepatic transplantation in the future. The pathophysiology of NAFLD is complex and involves multiple hits, but the principal contributing factor to its development is hepatic lipid accumulation, which leads to hepatic insulin resistance

Thyroid hormones are crucial in multiple physiological processes like homeostasis, mineral, lipid, carbohydrates, and protein metabolisms. Lipid metabolism has been reported, such as increased metabolic rate, weight loss, lipolysis, and lowering serum cholesterol levels. The physiological process of thyroid hormones (TH) affects almost every organ, and the liver is one of the most critical targets of TH.. Low thyroid hormone function may cause hypercholesterolemia which plays a fundamental role in the pathophysiology of hypothyroidism-induced NAFLD The prevalence of NAFLD among the population drastically increased in the last twenty years. NAFLD manifests itself in various ways in people worldwide, affecting both the female and male sex. The global prevalence of NAFLD is 25 percent, which is approximately as high as one billion and growing. One of the most common causes of chronic liver disease in the United States is NAFLD. It affects 80 to 100 million people, and approximately 25% of the cases progress to NASH. NAFLD includes a wide range of histopathological conditions such as non-alcoholic fatty liver (NAFL), non-alcoholic steatohepatitis (NASH), fibrosis, NASH cirrhosis, and NASH-related hepatocellular carcinoma (HCC). NAFLD is a diagnosis of exclusion. The number of NASH patients with cirrhosis is rising, resulting in an increase in liver transplantation for end-stage cirrhosis

. Accumulation of the lipids causes oxidative stress and inflammatory response in the liver . Another factor that may be involved in the thyroid-liver complex is leptin. Leptin is elevated in hypothyroid patients and is also elevated in NAFLD patients. Leptin can promote hepatic insulin resistance and play a role in hepatic fibrogenesis There is no drug therapy for hypothyroidism-induced NAFLD that is currently approved. Steatosis can be reduced through structured lifestyle changes such as weight loss, dietary changes such as reduced drinking of alcohol, decreasing intake of food and drinks that have a high level of fructose, and increased daily activities and workouts

ELIGIBILITY:
Inclusion Criteria:All cases of hypothyroidism -

Exclusion Criteria:Diabetic Patient , obesity grade 2

-

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypothyroidism patient
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
to estimate the percentage of NAFLD in patients of hypothyoidism | in about one year
  through performing abdominal ultrasound to at least 100 patients of hypothyoidism

CONTACTS AND LOCATIONS:
Overall Officials: wael ahmed abbas, prof, Study Director — Assiut University; walaa anwer shehata, prof, Study Director — Assiut University; mena sawerss fathy, residant, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanase DM, Gosav EM, Neculae E, Costea CF, Ciocoiu M, Hurjui LL, Tarniceriu CC, Floria M. Hypothyroidism-Induced Nonalcoholic Fatty Liver Disease (HIN): Mechanisms and Emerging Therapeutic Options. Int J Mol Sci. 2020 Aug 18;21(16):5927. doi: 10.3390/ijms21165927. PMID 32824723
- [Background] Kowalik MA, Columbano A, Perra A. Thyroid Hormones, Thyromimetics and Their Metabolites in the Treatment of Liver Disease. Front Endocrinol (Lausanne). 2018 Jul 10;9:382. doi: 10.3389/fendo.2018.00382. eCollection 2018. PMID 30042736
- [Background] Chung GE, Kim D, Kim W, Yim JY, Park MJ, Kim YJ, Yoon JH, Lee HS. Non-alcoholic fatty liver disease across the spectrum of hypothyroidism. J Hepatol. 2012 Jul;57(1):150-6. doi: 10.1016/j.jhep.2012.02.027. Epub 2012 Mar 14. PMID 22425701
- [Background] Perumpail BJ, Khan MA, Yoo ER, Cholankeril G, Kim D, Ahmed A. Clinical epidemiology and disease burden of nonalcoholic fatty liver disease. World J Gastroenterol. 2017 Dec 21;23(47):8263-8276. doi: 10.3748/wjg.v23.i47.8263. PMID 29307986
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Zhu B, Chan SL, Li J, Li K, Wu H, Cui K, Chen H. Non-alcoholic Steatohepatitis Pathogenesis, Diagnosis, and Treatment. Front Cardiovasc Med. 2021 Sep 7;8:742382. doi: 10.3389/fcvm.2021.742382. eCollection 2021. PMID 34557535
- [Background] Mandato C, D'Acunzo I, Vajro P. Thyroid dysfunction and its role as a risk factor for non-alcoholic fatty liver disease: What's new. Dig Liver Dis. 2018 Nov;50(11):1163-1165. doi: 10.1016/j.dld.2018.08.026. Epub 2018 Sep 1. No abstract available. PMID 30262159
- [Background] He W, An X, Li L, Shao X, Li Q, Yao Q, Zhang JA. Relationship between Hypothyroidism and Non-Alcoholic Fatty Liver Disease: A Systematic Review and Meta-analysis. Front Endocrinol (Lausanne). 2017 Nov 29;8:335. doi: 10.3389/fendo.2017.00335. eCollection 2017. PMID 29238323
- [Background] Sanyal D, Mukherjee P, Raychaudhuri M, Ghosh S, Mukherjee S, Chowdhury S. Profile of liver enzymes in non-alcoholic fatty liver disease in patients with impaired glucose tolerance and newly detected untreated type 2 diabetes. Indian J Endocrinol Metab. 2015 Sep-Oct;19(5):597-601. doi: 10.4103/2230-8210.163172. PMID 26425466
- [Background] Liebe R, Esposito I, Bock HH, Vom Dahl S, Stindt J, Baumann U, Luedde T, Keitel V. Diagnosis and management of secondary causes of steatohepatitis. J Hepatol. 2021 Jun;74(6):1455-1471. doi: 10.1016/j.jhep.2021.01.045. Epub 2021 Feb 10. PMID 33577920